CLINICAL TRIAL: NCT05502419
Title: Effects of Neural Slump Mobilization in Addition to Conventional Physical Therapy in Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2022/8
Record Dates: First submitted 2022-08-10; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial which will consist of two groups. Once will recieve conventional physcial therapy and the sencond will recieve conventional physcial therapy and slump stretching.Both groups will be recruited concurrently.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be a another person who will be unaware of the group the participant belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional physical therapy (Active Comparator)
  Interventions: Procedure: Conventional Physical Therapy
- conventional physical therapy with slump stretching (Experimental)
  Interventions: Procedure: Neural slump mobilization; Procedure: Conventional Physical Therapy

INTERVENTIONS:
Procedure: Neural slump mobilization — Slump stretching will be performed with the patient in the long sitting position with the patient's feet against the wall to assure the ankle remained in 0 degree dorsiflexion. The therapist will apply over pressure to the cervical spine flexion to the point where the patient's symptoms will be reproduced. The position will be held for 30 s. A total of 5 repetitions will be completed.
  Arms: conventional physical therapy with slump stretching
Procedure: Conventional Physical Therapy — Moist heat with hydro collator pack, Maitland Mobilization for Lumbar spine, Therapeutic exercise: Core stability exercises

SUMMARY:
Low back pain is amongst the most prevalent musculoskeletal conditions worldwide.This condition has a significant impact on the person's quality of life by effecting their various activities of daily living. As of 2017 it remains the leading cause of years lived with disability.Various management strategies are used for the treatment of low back pain. In the recent years neurodynamic techniques are being used for the treatment of low back pain. Escpecially, patients of low back pain who have neural mechanosensitivity may benefit from neural mobilization techniques. Slump stretching is a neurodynamic technqiue which is used to improve the mobility of dural tissue.Different studies have shown postive results of slump stretching in patients of low back pain. However no such study has investigated the role of slump stretching in improving range of motiion in low back pain patients.So this study aims to investigate the the effect of slump stretching in low back pain patients specially on low back Low back pain is amongst the most prevalent musculoskeletal conditions worldwide.This condition has a significant impact on the person's quality of life by effecting their various activities of daily living. As of 2017 it remains the leading cause of years lived with disability.Various management strategies are used for the treatment of low back pain. In the recent years neurodynamic techniques are being used for the treatment of low back pain. Escpecially, patients of low back pain who have neural mechanosensitivity may benefit from neural mobilization techniques. Slump stretching is a neurodynamic technqiue which is used to improve the mobility of dural tissue.Different studies have shown postive results of slump stretching in patients of low back pain. However no such study has investigated the role of slump stretching in improving range of motiion in low back pain patients.So this study aims to investigate the the effect of slump stretching in low back pain patients specially on low back

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-44 years
* Both males and females
* Persons with low back pain with a positive slump test
* Patients with a NPRS intensity of at least 5

Exclusion Criteria:

* Patients with signs or symptoms of nerve root involvement
* Pregnant females, patients with history of spinal surgery, patients of spondylolistheis, spinal stenosis and disc herniation.
* Patients with serious spinal conditions infection, tumors, osteoporosis, spinal fracture

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
ROM | 2 weeks
  Range of motion will be measured with gravity based inclinometer. One inclinometer will be placed on T12 spinous process and the second inclinometer will be placed on S1 spinous process of participant. The patient is asked to perform forward flexion, extension and lateral flexion, The range of motion is recorded by subtracting the value on lower inclinometer from upper inclinometer.

SECONDARY OUTCOMES:
Back Pain | 2 weeks
  Back Pain will be measured via Numeric Pain Rating Scale. A higher score will signify higher level of pain.
Physical Function | 2 weeks
  Repeated sit to stand test will be used to assess the physical function of the participant
Disability | 2 weeks
  Disability will be assessed via Pain Disability Index. A higher score signifies poor outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Fauji Foundation Hospital, Rawalpindi, Punjab Province, Pakistan